CLINICAL TRIAL: NCT02354287
Title: Effectiveness of Cold Biopsy Forceps With Pre-lift for Complete Resection of Colonic Polyps ≤7mm in Size.
Status: Completed | Type: Observational
Sponsor: Gloucestershire Hospitals NHS Foundation Trust (Other)
Collaborators: Olympus (Industry)
Responsible Party: Sponsor
Other Study IDs: 166725
Record Dates: First submitted 2015-01-13; First posted 2015-02-03 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Colorectal Polyps

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients having outpatient Colonoscopy.: Patients with Polyps ≤7mm that are deemed appropriate to be removed by cold forceps polypectomy with pre lift
  Interventions: Procedure: Cold forceps polypectomy with pre lift

INTERVENTIONS:
Procedure: Cold forceps polypectomy with pre lift — Polyps ≤7mm will be included in the study if deemed appropriate by the colonoscopist..
  These polyps will be resected with cold forceps after pre injection into the submucosa with a few millilitres of pre injection solution (19 ml gelofusine, 1ml 1:10000 adrenaline and 1ml indigo carmine). Polyps are grasped with the cold forceps and pulled away from the rest of the colonic mucosa. Attempt will be made to remove polyps with single attempt with the forceps however several grasps may be required for complete visual resection of the polyp.
  The polypectomy site and a 5mm rim of normal appearing tissue will then be resected with endomucosal resection (EMR) using conventional snare method. This is to ascertain if there is any residual polyp tissue.
  Other Names: polypectomy

SUMMARY:
There is no consensus method for removal of diminutive (5mm) to small(6-9mm) colorectal polyps at colonoscopy. Neither the European Society of Gastrointestinal Endoscopy or the American Society of Gastrointestinal Endoscopy have guidelines for the removal of these polyps, despite the fact that around 90% of lesions removed by polypectomy at colonoscopy are diminutive to small.

Multiple techniques are used for polyp removal, especially diminutive lesions. These include either forceps, both hot and cold, as well as snare with electrocautery or cold snare. Forceps utilises shearing force to grasp tissue and remove it, with the hot method passing a current through the grasper to essentially burn tissue. Snare is the use of a small metal loop placed and tightened at the base of polyps to cut through the tissue either straight away in a cold method or with electrocautery where a small current is passed through the loop to assist cutting through tissue. Surveys of Colonoscopists and Gastroenterologists in Australia and the United States show that the choice of method used for diminutive to small polyps is highly variable with cold snaring marginally favoured.Studies into polypectomy techniques are limited and it is clear that additional data and the review of polypectomy methods needs to be undertaken in order determine the optimal method for the removal of diminutive and small colorectal polyps.

A technique is used at the Gloucestershire National Health Service (NHS) trust involving a submucosal pre injection with a standard solution then the use of cold forceps for removal of polyps ≤7mm. This appears to be both very safe and highly effective method for the removal of these lesions compared to other techniques. No formal published studies have been completed to evaluate this method at national and international levels. We propose a study to evaluate the effectiveness, safety and costs of this method.

DETAILED DESCRIPTION:
Hypothesis A pre injection and cold forceps technique for removal of polyps ≤ 7mm is safe and results in retrieval rates >98% with complete histological resection >90% of the time.

Objectives

1. Determine the histological complete resection rate (CRR) using a pre injection lift and cold forceps for polypectomy of polyps ≤7mm.
2. Determine the number of bites required for complete visual resection of these polyps and the time taken from the beginning of pre injection needle insertion till complete resection.
3. To determine the polyp retrieval rate of this method.
4. To record any complications from this technique.
5. To compare the CRR, number of biopsies for visual eradication, time taken, polyp retrieval rate and complication rate of this method to cold forceps alone and cold snare from previous studies.

Methods

Participants:

Sample size 150 polyps, anticipated to be captured in between 75 and 100 patients based on an average of 2 polyps per patient. There is no published data on this polypectomy technique and there is limited data on other diminutive to small polypectomy techniques. Other comparative published studies looking at polypectomy techniques for diminutive to small polyps have had polyp numbers between fifty four and one hundred and seventeen.The sample size of 150 polyps is an approximation based on the fact that it is an achievable figure within the scope of the project and local clinical service which should yield a relatively narrow confidence interval.

Colonoscopists 3 experienced Gastroenterologists (JA, TB, PD) working within the Gloucestershire NHS Trust, each having performed over 3000 colonoscopies. All Gastroenterologists are certified British Bowel Cancer Screening Program Colonoscopists. As the technique being studied is already well practiced within the trust the extra time required for each polyp included in the study is negligible.

Pathologist All Polypectomy specimens and EMR tissue will be examined by an expert Gastrointestinal Pathologist (NS) who will be blinded to the patient and colonoscopist details when examining specimens.

The additional work for the pathology department is negligible. It can be routine practice to take additional material for analysis if incomplete removal of the polyp is suspect. In the study all polyps will have this review. NS will provide consistency and also time to support us in this project.

Course of Action:

1. Patients will be consented to participate in the study prior to their procedure. Information regarding the study will be posted to the patient at least a week prior to their colonoscopy.
2. If patient agrees to participate details including age, sex and indication for scope will be recorded. This data will be recorded with a patient study number. The patients will be otherwise anonymised.
3. Data from each colonoscopy and polypectomy will be recorded, including polyp size, location, time for resection, bites required for complete visual resection (another study showed the median number of bites to be at 2 with range 1-5 ), overall withdrawal time and quality of bowel preparation at the time of the procedure. Any adverse events at the time of colonoscopy, polypectomy and EMR or at subsequent patient follow up 7 days post procedure will be recorded prospectively on form A (Appendix 1) and also reported to the Research and Development team within 7 days of the Investigators becoming aware of the adverse event.

3. All colonoscopies will be performed using Olympus 240 and 260 colonoscopes with magnetic endoscopic imaging and Narrow band imaging (NBI) available to the Colonoscopist if required.

5. The equipment used for each polypectomy and Endomucosal resection (EMR) of polypectomy site will include the following.

1. Needle for pre injection
2. Pre injection mix will include 19 ml gelofusine, 1ml 1:10000 adrenaline and 1ml indigo carmine.
3. Cold forceps with span of 6.8mm and capacity of 7.22mm3
4. Olympus snare master 10mm snare.

   6. Any complications relating to the polypectomy will be recorded. 7. Polyps ≤7mm will be included in the study if deemed appropriate by the colonoscopist. Polyps may be considered inappropriate if polyp location or appearance is not suitable for the technique being studied.

   8. These polyps will be resected with cold forceps after pre injection into the submucosa. Data related to this resection will be recorded as noted above.

   9. The polypectomy site will then be resected with EMR using conventional snare method to ascertain if there is any residual polyp tissue. This is the only additional step to the polypectomy process which would not otherwise take place. The risk from this step of an adverse event to the patient would be significantly less than the risk of complication from a therapeutic Colonoscopy which is between 0.05 and 0.07%. A maximum of 3 polyps per patient will be included for study analysis in order to ensure both patient and colonoscopist time at procedure does not differ significantly from what it would normally.

   10. Both EMR specimen and resected polyp tissue will be sent for histopathological evaluation by single expert Gastrointestinal Histopathologist who has kindly agreed to review the extra EMR tissue in his own time.

   11. Recruited patients will be called one-week post colonoscopy to ensure they do not wish to withdraw from the study and they have had no concerns post their procedure.

   Adverse Events As mentioned above the risk of adverse events related to the polypectomy technique being studied or the EMR of residual tissue is minimal.

   All adverse events (or medical occurrence) will be recorded in data collection spreadsheets. Any events classified as 'serious adverse events' (SAE) will be reported to the Research and Development Unit (RSDU).

   The following criteria will be used to assess the relationship (causality) of the adverse event to the polypectomy technique and EMR performed
   1. None: - The adverse event is definitely not associated with the investigational technique being used.
   2. Possible: - A causal relationship is possible when the adverse event follows a reasonable temporal sequence from the application of the intervention, but could have been produced by the patient's clinical state or other modes of treatment being administered to the patient.
   3. Probable: - The causal relationship is probable when the adverse event follows a reasonable temporal sequence from the application of the investigational technique. This is likely if the adverse event cannot be explained by the known characteristics of the patient's clinical state

   Adverse events will be assessed by one of the investigators who are qualified Gastroenterologists and managed accordingly.

   The severity of adverse events will be recorded using the following criteria:
   1. Mild: - Symptom(s) barely noticeable to the patient or does not make the patient uncomfortable. The AE does not influence performance or functioning.

      Prescription drugs are not ordinarily needed for relief of symptom(s).
   2. Moderate: - Symptom(s) of a sufficient severity to make the patient uncomfortable or require endoscopic intervention or other treatments.
   3. Severe: - Symptom(s) of a sufficient severity to cause the patient severe discomfort requiring subsequent treatment or require major endoscopic intervention, hospitalisation or surgery.

   A serious adverse event (SAE) includes adverse events that result in death, require either inpatient hospitalization or the prolongation of hospitalization, are life threatening, result in a persistent or significant disability/incapacity. Other important medical events, based upon appropriate medical judgement, may be considered Serious Adverse Events if a trial participant's health is at risk and intervention is required to prevent an adverse outcome.

   Dr Alex di Mambro FRCP (Gloucestershire NHS Trust Gastroenterologist) will evaluate, report and assist in patient management should there be a SAE. In no other way has she been involved in study development or will she be involved during the course of the study.

   All reports of serious adverse events (SAE) will be recorded on the SAE form for this trial and forwarded immediately to the Research & Development Unit (RSDU). A copy of this form can be seen in the appendix 1. In the event of a SAE persisting greater then 24 hours another form will be submitted to the RSDU. Also, in the case of a persisting SAE the time of event resolution, patient death or discharge a subsequent form will be completed and submitted.

   Data recording and statistical analysis: All data will be recorded prospectively in a Microsoft excel spread sheet by the chief investigator (SO) and statistical analysis completed with SPSS version 16. Based on a target sample size of 150 polyps with 90% success rate the calculated 95% confidence interval will be 84.5-94.2%.

   Data storage: The collected data will be kept secure within the department of Gastroenterology and not shared with uninvolved persons. The data will be anonymised and the excel sheet the data is collected on will be password protected and not available to other individuals not involved with the study. All recorded data will be destroyed by the end of calendar year 2017 or once the anonymised results have been presented and published which is expected to be by the end of calendar year 2015.

   Results It is anticipated that results of this study will be completed for abstract submission for United European Gastroenterology Week by May 2015. This meeting will be held in Europe in October 2015. We will aim to publish this data in an international Endoscopic journal by late 2015. Results will be made available to our Bowel Cancer screening nurses who will be able to disseminate these results to various Bowel Cancer support groups.

   Funding

   Researchers and Time allocation The chief investigator has time (20hr/week) allocated into current Gloucestershire NHS Trust contract for education and development. Development of this study, data recording/entry and generation of an academic paper will all be undertaken in this time.

   Professor Neil Shepherd, Pathologist for this project has agreed to undertake the additional work of EMR tissue review in his own time.

   Additional time for colonoscopists will be for EMR of polypectomy site that is considered negligible in the course of a standard colonoscopy.

   Equipment As explained in the methods section minimal additional pieces of equipment are needed compared to the standard colonoscopy. Snares for EMR of polypectomy site will only be additional should a snare not have already been required for the removal of larger polyps during the course of the colonoscopy.

   Olympus will kindly provide the additional snares for the study. All other equipment such as pre injection solution, pre injection needle and cold forceps would normally be used in the course of colonoscopy and polypectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients from Cheltenham General Hospital and Royal Gloucestershire Hospitals that have been scheduled for colonoscopy through our outpatient clinics or inpatient consult service will be prospectively recruited prior to their Colonoscopy.

Exclusion Criteria:

* Patients will be excluded if:

  1. They are under the age of 18.
  2. They do not have capacity to consent for the Colonoscopy as determined at the time of procedural admission by the trained admitting endoscopy nurse. If a patient is deemed to lack capacity by the referring doctor or admitting nurse this will also be assessed by the colonoscopist. Both the colonoscopist and admitting nurses have been trained to assess capacity,that is whether a persons mind is affected at the time of the procedure in such a way that they are unable to make a decision. There are multiple reasons as to why an individuals brain or mind may be altered such as medications, mental illness or dementia.
  3. There is a history of Inflammatory Bowel Disease
  4. Identified coagulopathy with PT>1.4 or thrombocytopenia with Platelets <80 on any bloods collected within routine clinical practice within the past 4 weeks. This will not be an additional procedure and these bloods are routinely taken on patients where coagulopathy or thrombocytopenia is a concern such as patients on long term Warfarin or with chronic liver disease. These patients are identified by Endoscopy nursing staff in pre assessment work up. Routine haematology is not taken as part of a standard assessment for outpatient endoscopy.
  5. Taking dual anti platelet therapy or pharmacological anti coagulation.
  6. Bowel preparation is deemed poor by colonoscopist.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Residents from within Gloucestershire, United Kingdom whom have been referred for a Colonoscopy through either.
  1. Bowel cancer screening program or outpatient referral
  2. Outpatient clinics
  3. Inpatient referral
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2015-02; Primary Completion 2015-09-25 (Actual); Study Completion 2015-09-25 (Actual)

PRIMARY OUTCOMES:
Histological complete resection rate (CRR) using a pre injection lift and cold forceps for polypectomy of polyps ≤7mm. | Within one week of patients colonoscopy
  Gastrointestinal pathologist will assess histology of polyp resected then assess the polypectomy site rim that was resected at EMR for any evidence of residual polyp that was not visible to the colonoscopist.

SECONDARY OUTCOMES:
The number of bites required for complete visual resection of these polyps and the time taken from the beginning of pre injection needle insertion till complete resection. | intraoperative during colonoscopy and analysed within one month of last patient recruitment
  Researcher will record time from pre injection till end of visual eradication of polyp.

OTHER OUTCOMES:
The polyp retrieval rate of this method. | intraoperative during patient colonoscopy and analysed within one month of last patients recruitment.
  Complete polyp retrieval is if all polyp tissue is successfully retrieved at the time of colonoscopy. Occasionally tissue may be dislodged from forceps and be misplaced within colon fluid and residue.
Immediate or delayed complications from this technique. | intraoperative and after one week.
  Common complications of polypectomy include bleeding, both immediate and delayed. Immediate bleeds will occur at the time of the colonoscopy and will be considered significant if endoscopic therapy is required to treat. Delayed bleeds will usually be within a week of the index procedure and will present as per rectal bleeding or haematochezia. This will only be determined to be related to the procedure if a repeat colonoscopy is performed and the bleeding site is assessed to be from a polypectomy site included in the study. Perforation of the colon would usually be determined during the colonoscopy, often at the time of polypectomy at the polypectomy site. A delayed perforation is also possible usually within 48 hours of the procedure and is often determined with computer tomography (CT) scan.
An overall comparison of this polypectomy method compared to other methods used for diminutive and small polyps. | 2 months post completion of recruitment.
  A direct comparison of CRR, number of biopsies for visual eradication, time taken for procedure, polyp retrieval rate and complication rate to other techniques primarily cold snare and cold forceps without a pre-lift.

CONTACTS AND LOCATIONS:
Overall Officials: Sam A O'Connor, FRACP, Principal Investigator — Advanced Endoscopy and Gastroenterology Fellow
Locations (1):
- Cheltenham General Hospital, Cheltenham, Gloucestershire, United Kingdom

REFERENCES:
- [Background] Winawer SJ, Zauber AG, Ho MN, O'Brien MJ, Gottlieb LS, Sternberg SS, Waye JD, Schapiro M, Bond JH, Panish JF, et al. Prevention of colorectal cancer by colonoscopic polypectomy. The National Polyp Study Workgroup. N Engl J Med. 1993 Dec 30;329(27):1977-81. doi: 10.1056/NEJM199312303292701. PMID 8247072
- [Background] Zauber AG, Winawer SJ, O'Brien MJ, Lansdorp-Vogelaar I, van Ballegooijen M, Hankey BF, Shi W, Bond JH, Schapiro M, Panish JF, Stewart ET, Waye JD. Colonoscopic polypectomy and long-term prevention of colorectal-cancer deaths. N Engl J Med. 2012 Feb 23;366(8):687-96. doi: 10.1056/NEJMoa1100370. PMID 22356322
- [Background] Atkin WS, Cook CF, Cuzick J, Edwards R, Northover JM, Wardle J; UK Flexible Sigmoidoscopy Screening Trial Investigators. Single flexible sigmoidoscopy screening to prevent colorectal cancer: baseline findings of a UK multicentre randomised trial. Lancet. 2002 Apr 13;359(9314):1291-300. doi: 10.1016/S0140-6736(02)08268-5. PMID 11965274
- [Background] Farrar WD, Sawhney MS, Nelson DB, Lederle FA, Bond JH. Colorectal cancers found after a complete colonoscopy. Clin Gastroenterol Hepatol. 2006 Oct;4(10):1259-64. doi: 10.1016/j.cgh.2006.07.012. Epub 2006 Sep 25. PMID 16996804
- [Background] Martinez ME, Baron JA, Lieberman DA, Schatzkin A, Lanza E, Winawer SJ, Zauber AG, Jiang R, Ahnen DJ, Bond JH, Church TR, Robertson DJ, Smith-Warner SA, Jacobs ET, Alberts DS, Greenberg ER. A pooled analysis of advanced colorectal neoplasia diagnoses after colonoscopic polypectomy. Gastroenterology. 2009 Mar;136(3):832-41. doi: 10.1053/j.gastro.2008.12.007. Epub 2008 Dec 9. PMID 19171141
- [Background] Pabby A, Schoen RE, Weissfeld JL, Burt R, Kikendall JW, Lance P, Shike M, Lanza E, Schatzkin A. Analysis of colorectal cancer occurrence during surveillance colonoscopy in the dietary Polyp Prevention Trial. Gastrointest Endosc. 2005 Mar;61(3):385-91. doi: 10.1016/s0016-5107(04)02765-8. PMID 15758908
- [Background] Leung K, Pinsky P, Laiyemo AO, Lanza E, Schatzkin A, Schoen RE. Ongoing colorectal cancer risk despite surveillance colonoscopy: the Polyp Prevention Trial Continued Follow-up Study. Gastrointest Endosc. 2010 Jan;71(1):111-7. doi: 10.1016/j.gie.2009.05.010. Epub 2009 Jul 31. PMID 19647250
- [Background] Lieberman D, Moravec M, Holub J, Michaels L, Eisen G. Polyp size and advanced histology in patients undergoing colonoscopy screening: implications for CT colonography. Gastroenterology. 2008 Oct;135(4):1100-5. doi: 10.1053/j.gastro.2008.06.083. Epub 2008 Jul 3. PMID 18691580
- [Background] Regula J, Rupinski M, Kraszewska E, Polkowski M, Pachlewski J, Orlowska J, Nowacki MP, Butruk E. Colonoscopy in colorectal-cancer screening for detection of advanced neoplasia. N Engl J Med. 2006 Nov 2;355(18):1863-72. doi: 10.1056/NEJMoa054967. PMID 17079760
- [Background] Chandran S, Parker F, Vaughan R, Efthymiou M. The current practice standard for colonoscopy in Australia. Gastrointest Endosc. 2014 Mar;79(3):473-9. doi: 10.1016/j.gie.2013.10.050. Epub 2013 Dec 12. PMID 24332081
- [Background] Singh N, Harrison M, Rex DK. A survey of colonoscopic polypectomy practices among clinical gastroenterologists. Gastrointest Endosc. 2004 Sep;60(3):414-8. doi: 10.1016/s0016-5107(04)01808-5. PMID 15332033
- [Background] Repici A, Hassan C, Vitetta E, Ferrara E, Manes G, Gullotti G, Princiotta A, Dulbecco P, Gaffuri N, Bettoni E, Pagano N, Rando G, Strangio G, Carlino A, Romeo F, de Paula Pessoa Ferreira D, Zullo A, Ridola L, Malesci A. Safety of cold polypectomy for <10mm polyps at colonoscopy: a prospective multicenter study. Endoscopy. 2012 Jan;44(1):27-31. doi: 10.1055/s-0031-1291387. Epub 2011 Nov 28. PMID 22125197
- [Background] Lee CK, Shim JJ, Jang JY. Cold snare polypectomy vs. Cold forceps polypectomy using double-biopsy technique for removal of diminutive colorectal polyps: a prospective randomized study. Am J Gastroenterol. 2013 Oct;108(10):1593-600. doi: 10.1038/ajg.2013.302. Epub 2013 Sep 17. PMID 24042189
- [Background] Deenadayalu VP, Rex DK. Colon polyp retrieval after cold snaring. Gastrointest Endosc. 2005 Aug;62(2):253-6. doi: 10.1016/s0016-5107(05)00376-7. PMID 16046990
- [Background] Komeda Y, Suzuki N, Sarah M, Thomas-Gibson S, Vance M, Fraser C, Patel K, Saunders BP. Factors associated with failed polyp retrieval at screening colonoscopy. Gastrointest Endosc. 2013 Mar;77(3):395-400. doi: 10.1016/j.gie.2012.10.007. Epub 2012 Dec 1. PMID 23211749
- [Background] Efthymiou M, Taylor AC, Desmond PV, Allen PB, Chen RY. Biopsy forceps is inadequate for the resection of diminutive polyps. Endoscopy. 2011 Apr;43(4):312-6. doi: 10.1055/s-0030-1256086. Epub 2011 Mar 16. PMID 21412704
- [Background] Jung YS, Park JH, Kim HJ, Cho YK, Sohn CI, Jeon WK, Kim BI, Sohn JH, Park DI. Complete biopsy resection of diminutive polyps. Endoscopy. 2013 Dec;45(12):1024-9. doi: 10.1055/s-0033-1344394. Epub 2013 Aug 6. PMID 23921846
- [Background] Metz AJ, Moss A, McLeod D, Tran K, Godfrey C, Chandra A, Bourke MJ. A blinded comparison of the safety and efficacy of hot biopsy forceps electrocauterization and conventional snare polypectomy for diminutive colonic polypectomy in a porcine model. Gastrointest Endosc. 2013 Mar;77(3):484-90. doi: 10.1016/j.gie.2012.09.014. Epub 2012 Nov 27. PMID 23199650
- [Background] Buchner AM, Guarner-Argente C, Ginsberg GG. Outcomes of EMR of defiant colorectal lesions directed to an endoscopy referral center. Gastrointest Endosc. 2012 Aug;76(2):255-63. doi: 10.1016/j.gie.2012.02.060. Epub 2012 May 31. PMID 22657404
- [Background] Church JM. Experience in the endoscopic management of large colonic polyps. ANZ J Surg. 2003 Dec;73(12):988-95. doi: 10.1046/j.1445-2197.2003.t01-23-.x. PMID 14632888
- [Background] Ferrara F, Luigiano C, Ghersi S, Fabbri C, Bassi M, Landi P, Polifemo AM, Billi P, Cennamo V, Consolo P, Alibrandi A, D'Imperio N. Efficacy, safety and outcomes of 'inject and cut' endoscopic mucosal resection for large sessile and flat colorectal polyps. Digestion. 2010;82(4):213-20. doi: 10.1159/000284397. Epub 2010 Jun 24. PMID 20588036
- [Background] Moss A, Bourke MJ, Williams SJ, Hourigan LF, Brown G, Tam W, Singh R, Zanati S, Chen RY, Byth K. Endoscopic mucosal resection outcomes and prediction of submucosal cancer from advanced colonic mucosal neoplasia. Gastroenterology. 2011 Jun;140(7):1909-18. doi: 10.1053/j.gastro.2011.02.062. Epub 2011 Mar 8. PMID 21392504
- [Background] Ichise Y, Horiuchi A, Nakayama Y, Tanaka N. Prospective randomized comparison of cold snare polypectomy and conventional polypectomy for small colorectal polyps. Digestion. 2011;84(1):78-81. doi: 10.1159/000323959. Epub 2011 Apr 14. PMID 21494037
- [Background] Warren JL, Klabunde CN, Mariotto AB, Meekins A, Topor M, Brown ML, Ransohoff DF. Adverse events after outpatient colonoscopy in the Medicare population. Ann Intern Med. 2009 Jun 16;150(12):849-57, W152. doi: 10.7326/0003-4819-150-12-200906160-00008. PMID 19528563